CLINICAL TRIAL: NCT07301697
Title: Safety and Performance Profile of Cryobiopsy in Bronchial Endoscopy
Acronym: SeReCryo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 9624; 2025-A01681-48 (Other: ANSM)
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Mediastinal Lymphadenopathy; Mediastinal Lesions; Diffuse Interstitial Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients who underwent a cryobiopsy (Experimental): performing a transbronchial cryobiopsy or EBUS-cryobiopsy on a patient with an evaluation for diffuse interstitial lung disease
  Interventions: Diagnostic Test: performance of a transbronchial cryobiopsy or EBUS-cryobiopsy

INTERVENTIONS:
Diagnostic Test: performance of a transbronchial cryobiopsy or EBUS-cryobiopsy — Transbronchial cryobiopsy is a relatively recent technique that is increasingly used for the diagnosis of various respiratory pathologies, notably neoplasms, diffuse interstitial lung diseases (ILDs), and rejection after lung transplantation. Currently, its use is integrated into European recommendations for the diagnosis of interstitial lung diseases. EBUS-cryobiopsy, on the other hand, has proven useful in the exploration of lesions and mediastinal lymphadenopathies. Several studies have compared this method to the reference technique, EBUS-TBNA (endobronchial ultrasound-guided transbronchial needle aspiration), and the results suggest a superior diagnostic yield of cryobiopsy, particularly for the detection of benign lesions and lymphomas.

SUMMARY:
Transbronchial cryobiopsy is a relatively recent technique, increasingly used for the diagnosis of various respiratory diseases, including neoplasms, diffuse interstitial lung diseases (ILDs), and rejection after lung transplantation. Currently, its use is included in European recommendations for the diagnosis of interstitial lung diseases. EBUS-cryobiopsy, on the other hand, has proven useful in the evaluation of lesions and mediastinal lymphadenopathy. Several studies have compared this method to the reference technique, EBUS-TBNA (endobronchial ultrasound-guided transbronchial needle aspiration), and the results suggest a higher diagnostic yield for cryobiopsy, particularly for detecting benign lesions and lymphomas. However, to date, no French recommendation has yet been published regarding the precise role of this examination in the management of mediastinal lesions. Since July 2024, transbronchial cryobiopsies and EBUS-cryobiopsies have been routinely performed in the thoracic endoscopy department of Strasbourg University Hospital by an experienced team of interventional pulmonologists. The indications are those described above, after approval in a multidisciplinary consultation meeting. The number of prospective studies on cryobiopsies is currently limited. With this study, the investigators aim to carry out work intended to complement the current data on the profitability and safety of using cryobiopsies in the center, based on their results obtained since July 2024, as well as through prospective data collection from procedures performed over a one-year period. In addition to a prospective component, this study has the strong point of evaluating the procedure conducted by a limited number of experienced operators, thereby reducing the risk of significant inter-operator variability, as has been observed in previous studies. Finally, this is the first French study on the subject. The investigators hypothesize that performing cryobiopsies in a large university hospital by experienced operators allows for obtaining satisfactory diagnostic results under good safety conditions.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have undergone, or are eligible for, a cryobiopsy according to national or international recommendations, or after failure of a first diagnostic test followed by a collegial discussion regarding the indication for cryobiopsy.
* Procedure performed within the bronchial endoscopy department of the New Civil Hospital of the University Hospitals of Strasbourg.
* For diffuse interstitial lung diseases: decision to perform a transbronchial cryobiopsy after case review in a multidisciplinary consultation meeting for patients whose specific type of ILD could not be determined with thoracic imaging and biological tests alone, for patients not eligible for surgical lung biopsy (SLB) due to the severity of their respiratory condition, or as an alternative to SLB (according to the recommendations of the European Respiratory Society).
* For lymph node puncture (EBUS-cryobiopsy): after discussing the case in a multidisciplinary concentration meeting, in patients with a lesion and/or mediastinal adenopathy, as a second- or third-line procedure, following the diagnostic failure of bronchial fibroscopy and/or transbronchial needle aspiration guided by endobronchial ultrasound (EBUS-TBNA). For patients with a strong suspicion of lymphoma, EBUS-cryobiopsy can be performed as a first-line procedure in parallel with EBUS-TBNA (which is systematically performed during the same procedure) in order to reduce the diagnostic delay.
* For the retrospective analysis: all patients who underwent a cryobiopsy, and those who had a CT-guided lung biopsy for diagnostic assessment of an ILD or evaluation of suspected pulmonary neoplasm, since July 2024.

Exclusion Criteria:

* - Patients under 18 years of age.
* Pregnant or breastfeeding women.
* Patients under guardianship, curatorship, or legal protection.
* Patients at increased risk of bleeding: patients on anticoagulants not stopped for 24 hours, or on direct oral anticoagulants not stopped for 5 days, or with INR > 1.5 for patients on VKAs and heparin. Patients on dual antiplatelet therapy. Platelet count below 50 G/L.
* Saturation below 90% on oxygen therapy with a maximum allowable flow of 2 L/min.
* Pre-existing severe heart disease: unstable angina, myocardial infarction, decompensated heart failure.
* Known pulmonary hypertension with systolic pulmonary arterial pressure above 50 mmHg on transthoracic echocardiography.
* Inability to provide the subject with informed information (emergency situation, subject has difficulty understanding, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-04-09 (Estimated); Study Completion 2027-04-19 (Estimated)

PRIMARY OUTCOMES:
Assess the diagnostic performance of transbronchial cryobiopsy and EBUS cryobiopsy in both indications | immediately after the intervention
  Determination of the exact diagnosis of ILD for patients with diffuse interstitial pneumonia confirmation of the diagnosis of the lesion (pulmonary neoplasm, lymphoma, sarcoidosis, etc.) in patients with mediastinal lesions and mediastinal lymphadenopathy

CONTACTS AND LOCATIONS:
Overall Officials: Michele PORZIO, Doctor, Principal Investigator — Pulmonology Department - Nouvel Hôpital Civil - HUS
Locations (1):
- Pulmonology Department - NHC Strasbourg, Strasbourg, France